CLINICAL TRIAL: NCT00706147
Title: Phase II/III Randomized, Placebo-Controlled Trial of Arimoclomol in SOD1 Positive Familial Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Phase II/III Randomized, Placebo-controlled Trial of Arimoclomol in SOD1 Positive Familial Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael Benatar, Professor, Department of Neurology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20100758; 3517 (Other Grant/Funding Number: OOPD)
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Hereditary ALS; Hereditary neurological disease; Lou Gehrig's Disease; Motor Neuron Disease; Amyotrophic Lateral Sclerosis (ALS); Familial ALS; Neuromuscular disease; SOD1 mutation; Superoxide dismutase; SOD1 positive ALS; inherited ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases | interventions — arimoclomol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Arimoclomol

INTERVENTIONS:
Drug: Arimoclomol — Drug: Arimoclomol capsules given three times per day
  Other Names: Arimoclomol (BRX-345)
  Arms: 2
Drug: Placebo — Drug: Placebo capsules given three times per day
  Arms: 1

SUMMARY:
The purpose of this study will be to demonstrate the safety, tolerability, and efficacy of arimoclomol in subjects with SOD1 positive familial Amyotrophic Lateral Sclerosis (ALS). This type of ALS is HEREDITARY (runs in families), and at least one other person in the family must have had ALS.

Study hypotheses: Arimoclomol, taken at a dose of 200 mg three times daily will improve survival as defined by time to death, tracheostomy or permanent assisted ventilation. In addition, it will be safe and well tolerated in subjects with SOD1 positive familial ALS.

Funding Source - FDA-OOPD

DETAILED DESCRIPTION:
Using a seamless, adaptive, phase II/III design, the investigators will determine the safety and efficacy of arimoclomol in patients with SOD1 positive familial ALS. Both stage-1 and stage-2 are randomized, double-blind and placebo-controlled in a population of patients with rapidly progressive SOD1 positive familial ALS. Patients with ALS, a history of a relative affected with ALS (i.e. familial ALS) and the presence of a demonstrable mutation in the SOD1 gene that is known to be associated with rapidly progressive disease, will be eligible for inclusion in this study. Potentially eligible subjects will undergo screening via telephone and, if necessary, review of outside medical records. The intervention will continue for up to 12 months. In the event that a participant reaches a study endpoint (e.g. tracheostomy or permanently assisted ventilation) study drug will be terminated. Subjects who meet all eligibility criteria will travel a study site for final eligibility determination, baseline evaluation and will then be randomized 1:1 to receive either placebo or arimoclomol at a dose of 200 mg t.i.d. Participants will then be evaluated again in person at a study site at Month-2. Telephonic evaluations at Month-1, 3, 4, 5, 6, 8, and 10 will be performed in participants' homes. Safety and tolerability evaluations will be performed at each of these visits. Collection of blood samples for safety laboratory analyses and measurement of blood pressure, heart rate, respiratory rate, temperature and weight will be performed at Months-1, 3, 4, 5, 6, 8, and 10 in the participant's home by a representative of a medical monitoring company. A study coordinator may perform an in-person visit at Month-12, or this visit may occur telephonically. A final evaluation will be performed via telephone at Month-13 (30 days after the last dose of study medication).

ELIGIBILITY:
Inclusion Criteria:

* Type of ALS that is hereditary (runs in families) only.
* El Escorial criteria for familial ALS and a family history of a pathogenic mutation in a gene known to be associated with ALS, such as the SOD1 gene.
* Willingness to undergo genetic testing and to learn the results.
* Demonstrable mutation in the SOD1 gene that is reported to be associated with a rapid rate of disease progression (i.e. A4V, A4T, C6F, C6G, V7E, L8Q, G10V, G41S, H43R, H48Q, D90V, G93A, D101H, D101Y, L106V, I112M, I112T, R115G, L126X, G127X, A145T, V148G, V148I) or possibly associated with rapidly progressive disease (E21G, G37R, L38V, D76Y, L84F, L84V, N86S, D90A het, G93R, I104F, I113T, L144F, L144S).
* Age 18 years or older; male or female.
* Capable of providing informed consent and complying with trial procedures.
* Diagnosis within less than 9 months of the anticipated date of the baseline visit AND study participants' subjective evaluation that they expect their physical condition to permit travel to the study site for both the baseline and 2-month study visits.
* Women must not be able to become pregnant (e.g. post menopausal for at least one year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. Adequate contraception includes: oral contraception, implanted contraception, intrauterine device in place for at least 3 months, or barrier method in conjunction with spermicide.
* Women of childbearing potential must have a negative pregnancy test at screening visit and be non-lactating.
* Willing to remain on a stable dose of Riluzole or to remain off Riluzole for the duration of the trial.
* Identifiable local medical doctor to assist with urgent care of any medical complications that may arise.
* Absence of any of the exclusion criteria.

Exclusion Criteria:

* History of known sensitivity or intolerability to Arimoclomol or to any other related compound.
* Exposure to any investigational drug within 30 days of the screening visit.
* Presence of any of the following clinical conditions:

  * Substance abuse within the past year.
  * Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active infectious disease.
  * AIDS or AIDS-related complex.
  * Unstable psychiatric illness defined as psychosis (hallucinations or delusions), untreated major depression within 90 days of the screening visit.
  * Positive pregnancy test at screening visit.
* Screening laboratory values:

  * Creatinine greater than 1.5.
  * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST). greater than 3.0 times the upper limit of normal.
  * Total bilirubin greater than 2.0 times the upper limit of normal.
  * White blood cell (WBC) count less than 3,500/mm3.
  * Platelet concentration less than 100,000/ul.
  * Hematocrit level less than 33 for female or less than 35 for male.
* Female patients who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Time to death, tracheostomy or permanent assisted ventilation will be the primary outcome measure. | 12 months

SECONDARY OUTCOMES:
Rate of decline of ALSFRS-R (ALS functional rating scale-revised) over a period of up to 12 months. | 12 months
Disease progression as measured by the rate of decline of FEV6. | 12 months
Safety and tolerability of arimoclomol will be evaluated by using vital signs and weight, clinical laboratory measures, physical examination, report of adverse events, and the proportion of subjects completing the study on assigned treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MBChB, DPhil, Principal Investigator — University of Miami; Merit Cudkowicz, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Benatar M, Wuu J, Andersen PM, Atassi N, David W, Cudkowicz M, Schoenfeld D. Randomized, double-blind, placebo-controlled trial of arimoclomol in rapidly progressive SOD1 ALS. Neurology. 2018 Feb 13;90(7):e565-e574. doi: 10.1212/WNL.0000000000004960. Epub 2018 Jan 24. PMID 29367439